CLINICAL TRIAL: NCT06596421
Title: Effect of Abdominal Massage on Constipation After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Gamze ataman YILDIZ, Chief Researcher, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20220750
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Massage
Keywords: Cardiac surgery; abdominal massage; constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experiment (Experimental): abdominal massage
  Interventions: Other: abdominal massage
- control (No Intervention): no intervention

INTERVENTIONS:
Other: abdominal massage — abdominal massage
  Arms: experiment

SUMMARY:
Background and Aim: Although the incidence of gastrointestinal complications after cardiovascular surgery is reported to be rare, it has been reported that patients experience problems with constipation within the week after discharge. The presence of abdominal distension due to constipation after cardiac surgery may lead to prolonged wound healing, paralytic ileus and gastric dilatation. This study aimed to evaluate the effect of abdominal massage on constipation after cardiac surgery.

Methods: A prospective, randomised controlled quasi-experimental study was conducted in the cardiovascular surgery clinic of a public hospital between September 2022 and July 2023. A power analysis was performed to determine the sample size. A total of 130 patients were randomly assigned to the experimental or control group using a simple randomisation method. Data were collected using a 21-item form from the first day after surgery. Burping and defecation times of the patients were evaluated and recorded.

Results: The mean age of the experimental group was 55.2±13.3 years, while the mean age of the control group was 60.4±10.6 years (p=0.015). There was no statistically significant difference between the groups in terms of sociodemographic characteristics, bowel preparation and preoperative fasting times. It was observed that bowel sounds started earlier in the experimental group (70.8% on the first postoperative day) compared to the control group (46.2% on the first postoperative day) (X2=16.629; p=0.005). The first burping time measurements in the control group (x̄=46.415 hours) were higher than those in the experimental group (x̄=31.262 hours). Postoperative defecation time was longer in the control group (x̄=99.51 hours) than in the experimental group (x̄=61.611 hours).

ELIGIBILITY:
Inclusion Criteria:

* - Being older than 18 years
* Agreeing to participate in the study
* Undergoing a cardiac surgery
* Not having a barrier for communication
* Not having a mental or cognitive disability
* Not using constipation treatment (like laxatives or enemas)
* Having no history of constipation disorders or gastrointestinal surgery.

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
patient sociodemographic characteristics and physical measurements form | 2 days to 1 week
  It was noted how many hours after the operation he had intestinal gas.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir Universty, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No